CLINICAL TRIAL: NCT04215328
Title: Facilitated Release of Endogenous Enterokines: An Ambulatory Prospective Randomized Controlled Trial
Brief Title: Facilitated Release of Endogenous Enterokines
Acronym: F2G
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: Halyard Health (Industry); Wallace H. Coulter Foundation (Other)
Responsible Party: Principal Investigator, Elizabeth Beale, Assistant Professor, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: USC HS-13-00748
Record Dates: First submitted 2019-12-26; First posted 2020-01-02 (Actual); Last update posted 2020-01-07 (Actual); Status verified 2020-01

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Obesity; Diabetes Mellitus, Type 2; Nutrient
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mixed-Meal (Experimental): Ensure Nutrition Shake
  Interventions: Dietary Supplement: Mixed-Meal
- Electrolyte Solution (Placebo Comparator): Pedialyte Solution
  Interventions: Dietary Supplement: Electrolyte Solution

INTERVENTIONS:
Dietary Supplement: Mixed-Meal — Per 250ml bottle: 220 calories, protein 9g, carbohydrate 33g (15g sugar), fat 6g, sodium 190mg, potassium 390mg; 500mLs by tube daily in 4 doses
  Other Names: Ensure Nutrition Shake® (Abbott Park, Illinois, U.S.A.)
  Arms: Mixed-Meal
Dietary Supplement: Electrolyte Solution — Electrolyte Solution 500mLs by tube daily in 4 doses
  Other Names: Unflavored Pedialyte ® (Abbott Park, Illinois, U.S.A.)
  Arms: Electrolyte Solution

SUMMARY:
The overall objective is to develop therapy for obesity and diabetes that is as effective as gastric bypass surgery but without the cost and safety concerns.

DETAILED DESCRIPTION:
Gastric bypass leads to rapid, sustained diabetes remission in the majority of patients who undergo this procedure and is also highly effective therapy for obesity. However, currently <1% of medically-eligible patients undergo this or other bariatric operations due to cost and safety concerns. The approach is based on data suggesting that the benefit of gastric bypass is largely due to anatomical rearrangement of the intestine which leads to accelerated delivery of nutrients to the jejunum. This rerouting of nutrients stimulates the release of multiple neural, hormonal and enterokine responses that are associated with appetite suppression and improved glucose control. In this pilot proposal the question under investigation is whether repeated rapid delivery of a mixed meal directly to the jejunum can promote weight loss and glucose control.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes on oral antidiabetic medication
* BMI greater than or equal to 30kg/m2
* A1C less than 9%

Exclusion Criteria:

* Use of any of the following medications: dipeptide-peptidase IV (DPP-IV) inhibitors (e.g., sitagliptin), GLP-1 analogs (e.g., exenatide) or medication that could alter glucose tolerance (e.g. steroids)
* Contraindication to tube (e.g. Prior upper gastrointestinal bleed, or history of easy bleeding, altered foregut anatomy due to obstruction or surgery)
* Known cardiovascular disease other than controlled hypertension.
* Pregnancy or unwilling to take contraception
* Active esophagitis
* Known hiatal hernia
* Active gastric ulcer and/or duodenal ulcers,
* Previous restrictive surgery of the gastrointestinal tract
* Crohn's disease
* Active cancer
* History of gastrointestinal hemorrhage
* Known upper gastrointestinal lesions with potential to bleed
* Use of NSAIDs or anticoagulants
* Psychiatric disorders other than mild depression
* Likely inability to adhere to study protocol including alcohol or drug dependent patients
* Type I diabetes,
* Liver, kidney or multi-organ dysfunction.
* Known eating disorders
* Inability to attend scheduled or unanticipated study visits
* Known prior abdominal problems or operations that could lead to adhesions or strictures and that could prevent the spontaneous passage of a 10 French jejunal tube if it were to dislodge distally.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2014-11-01 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
Weight change between groups | Day 0 to Day 14
  Weight measured in kilograms taken before and immediately following the intervention period between the intervention and control group

SECONDARY OUTCOMES:
Caloric intake within and between groups | Day 0 to Day 14
  Caloric intake measured in kcal. Determined by consumption of provided food.
Weight change within group | Day 0 to Day 14
  Weight measured in kilgrams. Within group
Change in waist and hip measurements | Day 0 to Day 14
  Measured in centimeters. Between groups.
Change in systolic and diastolic blood pressure | Day 0 to Day 14
  Measured in mmHg for both. Between groups.
Change in heart rate | Day 0 to Day 14
  Measured in beats per minute. Between groups.
Changes in gut hormone levels | Day 0 to Day 14
  Including GLP-1, PYY, CCK, C-peptide, and insulin. Between groups.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Beale, MD, Principal Investigator — University of Southern California, Keck School of Medicine
Locations (1):
- Roybal Diabetes Management Clinic, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Beale EO, Lee W, Lee A, Lee C, Soffer E, Crookes PF, Eagilen K, Chen R, Mack WJ, Tong H. Effect of bolus enteral tube feeding on body weight in ambulatory adults with obesity and type 2 diabetes: a feasibility pilot randomized trial. Nutr Diabetes. 2020 Jun 17;10(1):22. doi: 10.1038/s41387-020-0125-6. PMID 32555148

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-03-11): https://cdn.clinicaltrials.gov/large-docs/28/NCT04215328/Prot_SAP_000.pdf